CLINICAL TRIAL: NCT04383990
Title: Comparison of Early Versus Late Administration of Insulin Glargine in Patients With type1 Diabetes During Fasting Ramadan
Brief Title: Early Versus Late Administration of Insulin Glargine in T1DM During Fasting Ramadan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJ19/175/J
Record Dates: First submitted 2020-04-14; First posted 2020-05-12 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2020-05

CONDITIONS: Type1diabetes; Fasting; Insulin
Keywords: Type1 Diabetes; Fasting; Insulin Glargine; Ramadan; Hypoglycemia
MeSH Terms: conditions — Fasting; Insulin Resistance; Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Open label Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Glargine (Active Comparator): To take insulin Glargine at 6-7 pm
  Interventions: Other: Timing of taking insulin
- Late Glargine (Active Comparator): To take insulin Glargine at 10-12 pm
  Interventions: Other: Timing of taking insulin

INTERVENTIONS:
Other: Timing of taking insulin — To take insulin Glargine early (6-7pm) or late (bedtime-10-12pm)

SUMMARY:
To compare different timing of insulin Glargine administration (early-6 pm versus standard bedtime-10 pm) as part of standard of care in patients with type1 diabetes who wish to fast the month of Ramadan.

DETAILED DESCRIPTION:
The investigators aim to compare the effectiveness and safety of two management strategies currently used in basal insulin adjustment for treatment of Type1 diabetes (T1DM) during fasting the holy month of Ramadan.

Primary Objective:

To determine if taking basal insulin Glargine at 6 pm is associated with less rates of hypoglycemia -(we will consider glucose level of 70 mg/dl ( 3.9 mmol/l) and below as the level of hypoglycemia ) - compared to bedtime timing (10-12pm) during fasting Ramadan in patients with T1DM

Secondary Objectives:

1. To estimate the difference between the two groups in glucose variability
2. To estimate the difference between the two groups in number of days they needed to brake their fast
3. To assess the difference in glycemic control between the two groups
4. To estimate the difference between the two groups in overnight and daytime hyperglycemia.
5. To estimate the difference between the two groups in rate of severe hyperglycemia and /or DKA

It is a multi-center open label randomized study that will take place in the diabetes/Endocrine clinics at National Guards Hospitals in four cities (Jeddah, Riyadh, Alhasa, and Dammam)

Variables to be Assessed:

1. Patient's demographics including (age, gender, type and duration of diabetes), and baseline measurements (weight, height,BMI, …).
2. Rate of Hypoglycemic events (as per SMBG records and CGM) in both groups
3. Number of days fasting was broken in both groups
4. Rate of severe hyperglycemic episodes (BG>250mg/dl) or DKA in both groups
5. Mean blood glucose for the month of Ramadan as calculated from sum of each patient's 7-point blood sugar home measurements in both groups.
6. Mean 24-hour blood glucose as measured by a continuous glucose monitoring devise in both groups.
7. Mean fasting blood glucose for the month period as calculated from patients home blood sugar measurements in both groups.
8. Mean 2-hour post-prandial blood glucose for the as calculated from patients home blood sugar measurements in both groups.
9. Fructosamine and HbA1c level before and after Ramadan in both groups

Results of this study will help fill a current gap of knowledge and may also contribute to the development of future guidelines for the management of type1DM during Ramadan.

ELIGIBILITY:
Inclusion Criteria:

1. DM type 1
2. Age > 14 years
3. Diagnosis of type 1 DM of more than 6 months.
4. Committed to do SMBG

Exclusion Criteria:

1. Renal and hepatic impairment
2. Adrenal insufficiency
3. Pregnancy
4. Alcohol consumption
5. Any diagnosed psychiatric disease

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Hypoglycemia incidence | Through study completion, an average of 3 months
  To determine if taking basal insulin Glargine at 6 pm is associated with less rates of hypoglycemia -(we will consider glucose level of 70 mg/dl ( 3.9 mmol/l) and below as the level of hypoglycemia ) - compared to bedtime timing (10-12pm) during fasting Ramadan in patients with T1DM.

SECONDARY OUTCOMES:
Glucose variability | Through study completion, an average of 3 months
  To estimate the difference between the two groups in glucose variability as measured by standard deviation on glucose monitoring
Days fast broken | Through study completion, an average of 3 months
  To estimate the difference between the two groups in number of days they needed to brake their fast
Glycemic control | Through study completion, an average of 3 months
  To assess the difference in glycemic control between the two groups as measured by hbA1c and frucosamine before and after Ramadan
Hyperglycemia | Through study completion, an average of 3 months
  To estimate the difference between the two groups in overnight and daytime rates of hyperglycemia (BG > 250 mg/dl)
Acute diabetes complications | Through study completion, an average of 3 months
  To estimate the difference between the two groups in rate of severe hyperglycemia (hypoglycemia associated with need for outside assisstance) and /or presentation to ER with Diabetic Keto-acidosis (DKA)

CONTACTS AND LOCATIONS:
Locations (1):
- KingAbullahIMRC, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided